CLINICAL TRIAL: NCT06281821
Title: Alcohol Use and Chronic Pain in Primary Care
Brief Title: Mobile App-based Approach for Reducing Pain and Hazardous Drinking: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Tibor Palfai, Professor of Psychological and Brain Sciences, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4947 [Study 2]
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Drinking; Chronic Pain
MeSH Terms: conditions — Alcohol Drinking; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Compare an intervention to an assessment only control condition
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor at follow-up timepoint is masked to condition. Baseline assessment occurs prior to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile App Intervention (Experimental): Mobile health intervention delivered through an app
  Interventions: Behavioral: mhealth-pc
- Control (No Intervention): Assessment Only Control condition

INTERVENTIONS:
Behavioral: mhealth-pc — Participants meet with an interventionist who explains the rationale for the mobile app. They complete video and survey-based intervention content each week for 8 weeks. App-based sessions are supplemented with brief chat-based coaching weekly.
  Arms: Mobile App Intervention

SUMMARY:
Chronic pain and heavy drinking are common co-occurring conditions among patients presenting to primary care settings. Given their impact on functioning and medical outcomes, there would be considerable benefit to developing an accessible, easily utilized, integrative approach to reduce alcohol use and pain that can be readily incorporated into the health care settings. The objective of this study is to test a modified version of a smartphone-based intervention for reducing pain and alcohol use among individuals experiencing chronic pain who engage in heavy drinking. The primary goal is to test the feasibility and acceptability of implementing this intervention in a sample that includes participants from rural areas and providing initial data on the utility of the intervention.

DETAILED DESCRIPTION:
Heavy alcohol use represents a significant risk for morbidity and mortality. Unfortunately, addressing unhealthy patterns of alcohol use is often a challenge as patients typically present to health care settings with co-morbid conditions that: (1) may make unhealthy drinking a lower priority health issue and (2) may impact the capacity for sustained alcohol-related change. Chronic pain is among the most common of these conditions. Pain is a frequent source of distress and disability and is one of the most frequent causes for health care visits. Pain is also an important trigger for alcohol use among patients who drink and is associated with the experience of negative alcohol-related consequences and unhealthy drinking over time. The experience of pain has also been shown to be associated with poorer responses to alcohol interventions. There are a number of challenges when attempting to treat co-occurring unhealthy drinking and pain among their patients. Pain management and reduction of alcohol use among those who engage in heavy alcohol use is often not adequately achieved with pharmacological treatments nor are pharmacological treatments indicated for common pain conditions. Moreover, despite the availability of evidence-based psychosocial interventions for unhealthy drinking and chronic pain, patients with each of these conditions typically show poor adherence to treatment. Given the rates of pain and unhealthy alcohol use and their impact on functioning and medical outcomes, there would be considerable benefit to an accessible, easily utilized, integrative approach to treat heavy alcohol use and pain that can be readily incorporated into health care settings. The objectives of this study are to test the acceptability and feasibility of a smartphone-based intervention for reducing pain and alcohol use among individuals who experience chronic pain and heavy drinking. In addition, the study will provide a preliminary effect size estimates of the intervention on outcomes.

ELIGIBILITY:
Inclusion Criteria

* 1 Heavy drinking by NIAAA guidelines (weekly limits [> 7 standard drinks for women or men age 65+, > 14 for men younger than 65], and/or a heavy drinking episode in the past month [>3 for women or men age 65+, > 4 for men younger than 65]) or by a positive USAUDIT-C score
* 2 Chronic pain [at least 3 months in duration] of at least moderate severity (4 or greater on the Numerical Pain Rating Scale from 0-10)

Exclusion Criteria:

* 1 If on medication for pain or alcohol, not on same dose for at least 2 months [Note: Participants who are on psychoactive medications for pain management may be included if they have a stable (at least 2 months) medication dose and state a willingness to continue use of medication as prescribed by their physician through the intervention phase]
* 2 Patients with bipolar disorder, schizophrenia, other psychotic disorder, or current suicidal intent.
* 3 Prior history of withdrawal-related seizures or delirium tremens
* 4 Current non-pharmacological treatment for alcohol use disorder or chronic pain.
* 5 Any acute life-threatening illness that requires treatment or intend to have surgery for a pain-related condition in the next 6-months
* 6 Pain that is related to a current cancer diagnosis
* 7 Patients who are unable to provide one or more individuals who will likely know where they are at follow up
* 8 Individuals who do not have a smartphone with which they can use to complete the remote study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Pain (average weekly), Enjoyment of Life, General Activity (PEG) Scale | 7-days
  Three items with 0-10 scales to assess chronic pain based on the dimensions of pain severity, impact on enjoyment in life, and interference with activity. Range 0-30. Higher scores reflect worse outcomes
Time Line Follow-Back-30 Day Weekly Drinking | past 30 days
  Average number of drinks per week over the past 30 days. Higher scores reflect worse outcomes.

SECONDARY OUTCOMES:
Time Line Follow-Back 30-Day Heavy Episodic Drinking | past 30 days
  number of heavy drinking episodes (for men 5 or more on single occasion for women 4+) over tha past 30 days. Higher values reflect worse outcomes
Perceptions of Treatment Questionnaire | Current perception of intervention assessed 12 weeks following baseline (4 weeks following intervention completion)
  Ratings of intervention satisfaction using Likert-scale items 0 "not at all" to 8 "very much" to assess degree of perceived help with pain and alcohol use, perceived helpfulness of intervention components. Higher scores reflect better outcomes
Systems Usability Scale | Current perception of intervention assessed 12 weeks following baseline (4 weeks following intervention completion)
  Three item Likert scale (scored 1 "strongly disagree' to 5 "strongly agree') to assess ease, speed of learning, confidence using the mobile app. Higher scores reflect better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States